CLINICAL TRIAL: NCT03942419
Title: A Multicenter, Double-Masked, Randomized, Placebo-Controlled Phase 3 Study of the Safety and Efficacy of Atropine 0.1% and 0.01% Ophthalmic Solutions Administered With a Microdose Dispenser for the Reduction of Pediatric Myopia Progression (The CHAPERONE Study)
Brief Title: Microdosed Atropine 0.1% and 0.01% Ophthalmic Solutions for Reduction of Pediatric Myopia Progression
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim Analysis reviewed by Data Monitoring Committee indicated futility
Sponsor: Eyenovia Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EYN-MYO-AT-31
Record Dates: First submitted 2019-05-07; First posted 2019-05-08 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Atropine; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: This is a multi-center, double masked, randomized, placebo-controlled study evaluating the efficacy of microdosed atropine 0.01%, atropine 0.1% and placebo ophthalmic solutions. Subjects will administer their assigned medication daily in both eyes for 36 months, then be re-randomized to the same or an alternative treatment arm and followed for an additional 12 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: There will be no differences in the presentation of study drug administered. All study personnel conducting ophthalmic assessments will be masked to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Atropine 0.1% Ophthalmic Solution (Experimental): Atropine 0.1% ophthalmic solution administered daily in both eyes using a microdose dispenser
  Interventions: Drug: Atropine 0.1% Ophthalmic Solution
- Atropine 0.01% Ophthalmic Solution (Experimental): Atropine 0.01% ophthalmic solution administered daily in both eyes using a microdose dispenser
  Interventions: Drug: Atropine 0.01% Ophthalmic Solution
- Placebo Ophthalmic Solution (Placebo Comparator): Placebo ophthalmic solution administered daily in both eyes using a microdose dispenser
  Interventions: Drug: Placebo Ophthalmic Solution

INTERVENTIONS:
Drug: Atropine 0.1% Ophthalmic Solution — Atropine 0.1% ophthalmic solution administered with a microdose dispenser
  Arms: Atropine 0.1% Ophthalmic Solution
Drug: Atropine 0.01% Ophthalmic Solution — Atropine 0.01% ophthalmic solution administered with a microdose dispenser
  Arms: Atropine 0.01% Ophthalmic Solution
Drug: Placebo Ophthalmic Solution — Placebo ophthalmic solution administered with a microdose dispenser
  Arms: Placebo Ophthalmic Solution

SUMMARY:
This study evaluates the progression of myopia in participants using microdosed atropine 0.01%, atropine 0.1%, or placebo ophthalmic solution. Eligible subjects will administer study medication daily in each eye for 48 months. Efficacy and safety assessments will be performed at visits scheduled for 1, 6, 12, 18, 24, 30 and 36 months after initiation of medication use. Subjects will be re-randomized at the 36 month visit, then followed at 6 month intervals for an additional year.

DETAILED DESCRIPTION:
Subjects will be evaluated for eligibility during an initial Screening Visit and enrolled after signing the study-specific informed consent form(s). Eligible subjects must complete a run-in period where they use the microdose dispenser to administer study drug "vehicle" solution daily in both eyes. After run-in, subjects return for a Baseline Visit and additional study eligibility assessments. Subjects who continue to be eligible will be equally randomized to one of the following treatment groups:

* Microdose atropine 0.1% ophthalmic solution
* Microdose atropine 0.01% ophthalmic solution
* Microdose placebo ophthalmic solution

Randomization will be stratified by iris color (e.g., dark and light) and study site. Study enrollment will be limited to a maximum of 50% of subjects who self-identify as East Asian ethnicity. Subjects will use their assigned study medication daily in both eyes and return for efficacy and safety assessments at 1, 6, 12, 18, 24, 30, and 36 months.

At the Month 36 Visit, subjects in the 2 atropine dose arms will be re-randomized to either placebo or 1 of the 2 doses of atropine ophthalmic solution, while subjects originally assigned to placebo will be re-randomized to one of the 2 atropine ophthalmic solution arms. After re-randomization, all subjects will be followed for an additional year with efficacy and safety examinations at Months 42 and 48.

ELIGIBILITY:
Inclusion Criteria:

* Refractive error by cycloplegic autorefraction: myopia -1.00 D to -6.00 D in both eyes; astigmatism ≤ 1.50 D in both eyes; anisometropia < 1.50 D.
* Best-corrected distance visual acuity in current correction of 0.2 logMAR or better with interocular difference ≤ 0.1 logMAR.
* Refractive correction for each eye meets the following criteria: myopia within ± 0.50 D of the manifest refraction at the Screening Visit; cylinder power within ± 0.50 D of the manifest refraction at the Screening Visit; when cylinder power is < 1.00 D, axis within ± 15 degrees of the manifest refraction; when cylinder power is ≥ 1.00 D, axis within ± 5 degrees of the manifest refraction.

Exclusion Criteria:

* Current or previous myopia treatment with non-study atropine, pirenzepine or other topical anti-muscarinic agent.
* Current use of bifocals, progressive-addition lenses, or multifocal soft contact lenses.
* Use of rigid gas permeable lenses, including orthokeratology lenses within 90 days of Screening.
* Known atropine allergy.
* Abnormality of the cornea, lens, central retina, iris or ciliary body.
* Current or prior history of manifest strabismus, amblyopia, or nystagmus.
* Prior eyelid, strabismus, intraocular, or refractive surgery.
* Intraocular pressure > 26 mmHg.
* History of premature birth by parent's report.
* Inability to perform protocol-prescribed testing due to preexisting neurological diagnoses, genetic syndrome, or other issues.
* Medical conditions predisposing patient to degenerative myopia, abnormal ocular refractive anatomy, and/or any history of intraocular surgery.
* Any systemic disease or condition that may affect visual function or development such as diabetes mellitus.
* Any ocular inflammation or external ocular inflammation within 30 days of Screening.
* History of punctal occlusion.
* Heterochromia.
* Lid squeezers.
* Participation in any study of an investigational, interventional product within 30 days prior to Screening Visit.
* Immediate family member of study staff designed to perform study evaluations or procedures.
* Pregnancy, or if sexually active, unwillingness to use an acceptable form of contraception during the study.
* Presence of a severe/serious ocular condition or any other unstable medical condition that, in the Investigator's opinion, may preclude study treatment or follow-up.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 438 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Myopia progression | 36 Months
  The proportion of primary study eyes showing less than 0.50 D (spherical equivalent) myopia progression compared to baseline measured using cycloplegic autorefraction.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - University of Alabama at Birmingham School of Optometry, Birmingham, Alabama
  - Midwestern University, Glendale, Arizona
  - Canyon City Eyecare, Azusa, California
  - UC Berkeley, Berkeley, California
  - Marshall Ketchum University College of Optometry, Los Angeles, California
  - Ratner Children's Eye Center, San Diego, California
  - Illinois College of Optometry, Chicago, Illinois
  - Midwestern University, Downers Grove, Illinois
  - SUNY College of Optometry, New York, New York
  - Wake Forest Health Network Ophthalmology - Oak Hollow, High Point, North Carolina
  - Oculus Research, Raleigh, North Carolina
  - The Ohio State University - College of Optometry, Columbus, Ohio
  - Scott & Christie and Associates, Cranberry Township, Pennsylvania
  - Salus University - The Eye Institute, Philadelphia, Pennsylvania
  - Primary Eyecare Group, Brentwood, Tennessee
  - Southern College of Optometry, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Virginia Pediatric Eye Center, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No